CLINICAL TRIAL: NCT03873441
Title: Innovative Game-Aided Rehabilitation Platform for Rehabilitation of Balance in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Collaborators: SDM College of Medical Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS22614 (H2019:081)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Balance; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer Games-Aided Balance Training Group (Experimental): The participants in CGR group will be asked to sit or stand (as per the screening result) on fixed & compliant surfaces; to use objects instrumented with the miniature motion mouse to play various therapeutic yet entertaining games while handling and moving the test therapeutic objects using bi-manual grip gradually progressing to head rotations (mouse mounted on a cap worn by participant); finally using trunk movements as a part of experimental therapy protocol. While performing CGR; children will be standing on a thin pressure mat (placed over fixed or compliant surface). This will allow us to record the information of COP displacement [body sway] while CGR intervention implementation. This information will be used to quantify therapy dosage. The CGR Group will receive a 45-60 minutes of session thrice a week for 12 weeks.
  Interventions: Other: Computer Games-Aided Balance Training Protocol
- Conventional Balance Training Group (Active Comparator): The control group will be receiving the conventional balance training for static and dynamic balance function improvement. The therapy will be provided in sitting or standing (as per the screening result) in a graded manner progressing from fixed surfaces to movable compliant surfaces. The Conventional Balance Training Group will receive a 45-60 minutes of session thrice a week for 12 weeks.
  Interventions: Other: Conventional Balance Training Protocol

INTERVENTIONS:
Other: Computer Games-Aided Balance Training Protocol — 1) Sitting Balance exercises while playing the interactive computer games starting with bi manual object placed in hands for controlling the games, then using the head rotation movements to control the games progressing to use of trunk motions to control games while balancing on the compliant surfaces in order to progress by increasing the balance costs.
  (2) Standing Balance exercises progressing from a fixed support surface to uneven, compliant surfaces like progression from standing over ground to sponge to air bladder as child tolerates increased balance costs.
  (3) Progression then to balancing while performing the visuomotor and visuospatial game tasks such as playing the games starting with bi-manual object placed in hands for controlling the games, then using the head rotation movements to control the games and then progressing to use of trunk motions to control games while balancing on compliant surface.
  (4) Progression to single-leg stance and stepping activities.
  Other Names: CGR Balance Training Protocol
  Arms: Computer Games-Aided Balance Training Group
Other: Conventional Balance Training Protocol — The following is a summary of the conventional physical therapy balance training protocol:
  1. Active-assisted stretching exercises for lower limb musculature focusing on postural control and improvement in dynamic stability,
  2. Balance and weight bearing exercises with multi-directional reach outs associated with trunk movements on fixed surface gradually progressing to unstable movable and compliant surfaces,
  3. Weight transfer exercises with multi-directional reach outs and
  4. Stepping exercises in different directions on variety of surfaces.
  Arms: Conventional Balance Training Group

SUMMARY:
The research project focuses on the evaluation of an engaging computer game-aided rehabilitation platform for use in rehabilitation of young children with cerebral palsy. The goal of this research program is to produce high quality therapeutic point-of-care approaches and cost-effective delivery systems leading to better long-term health outcomes. At present, the challenges entailed in providing therapy services continue to put identified children at risk of missing opportunities to maximize the neurodevelopmental capacities, sustain any behavioral recovery and prevent future complications.The program is grounded on the technological developments and on current research documenting the benefits of computer-aided learning tools, exercise gaming applications in rehabilitation and principles of adaptive learning and neuroplasticity. A randomized controlled trial (RCT) will be conducted to study the feasibility and effectiveness of a computer game-aided rehabilitation platform (CGR) for a repetitive task practice (RTP) protocol designed for training of balance in young children with Cerebral Palsy (CP).

DETAILED DESCRIPTION:
The research project focuses on the evaluation of an innovative, engaging computer game-aided rehabilitation platform for use in rehabilitation of young children with cerebral palsy. The goal of this research program is to produce high quality therapeutic point-of-care approaches and cost-effective delivery systems leading to better long-term health outcomes. At present, the challenges entailed in providing therapy services continue to put identified children at risk of missing opportunities to maximize the neurodevelopmental capacities, sustain any behavioral recovery and prevent future complications.

Canada and India face a growing population of children with neurodevelopmental disabilities distributed across broad geographic regions. Cerebral palsy (CP) is the most common neurodevelopmental disability in childhood. The prevalence of CP in developing countries is estimated to be 5 to 10 times greater than in North America. Children with CP face a substantial amount of balance impairments which results in limitations of the mobility functions necessary for activities of daily living. The ability to perform functional tasks in sitting and standing while maintaining the balance is an important predictor of success in daily activities and participation in school, leisure and other aspects of community life.

There are many things to consider when developing therapy programs designed to improve dynamic balance skills for these affected children to maximize the neurodevelopmental capacities and to prevent the development of secondary disabilities. Intense repetitive task practice (RTP) such as, constraint-induced movement therapy is one of the few effective neuro-rehabilitative strategies shown to improve motor function in children with CP, with potential to overcome developmental difficulties. Constraint induced movement therapy consists of constraining the use of the unaffected limb to encourage use of the affected limb. However it is often difficult to engage children in therapy and sustain motivation to engage in intense RTP and achieve the therapy goals. Thus, there is a need for effective approaches and tools that motivate young children with CP to complete long-term neuro-rehabilitation programs and to provide developmental opportunities.

Digital media and gaming have received considerable interest from researchers and clinicians as a model for learning a broad range of complex tasks and facilitating the transfer of skills to daily life. These emerging rehabilitation technologies have the potential to improve clinical outcomes and child participation because these are engaging, motivating and now accessible. For this purpose a computer game-aided rehabilitation platform (CRP) has been developed. This approach combines motor exercises with fun games appropriate for children with neuro- developmental disorders. The approach is designed to provide engaging, high-quality, personalized therapy in the clinical rehabilitation setting.

Research Goal:

This research project focuses on the evaluation of an engaging exercise computer game-aided platform and embedded assessment tools for use in clinical practice. The program is grounded on the technological developments and on current research documenting the benefits of computer-aided learning tools, exercise gaming applications in rehabilitation and principles of adaptive learning and neuroplasticity. A pilot study to examine the feasibility and benefits of a computer-aided, game-aided repetitive task practice (RTP) program designed for training of dynamic balance skills in young children with CP will be conducted.

RESEARCH PROJECT OBJECTIVE 1

The CGR includes a designed rehabilitation assessment game which is capable of monitoring every child's performance during therapy. It quantifies motor skill parameters, as well as, visual-spatial skills and executive cognitive functions. It produces electronic records for these outcome measures and thus allows us to track change over time. It also provides timely feedback to child, parents and the therapist.

Objective: To evaluate the test-retest reliability and convergent validity of the assessment tool embedded in the game-aided rehabilitation platform. Specifically for dynamic balance in children aged 3-8 years (n= 50) diagnosed with CP. The new tool will be compared to commonly used outcome measures i.e. Peabody Developmental Motor Scale version 2 (PDMS-2) and Gross Motor Function Measure (GMFM). This will provide a reliable test protocol and valid measures that can accurately and quickly quantify dynamic balance control function independent of object-task type, for use in daily clinical practice and research. It is hypothesized that the performance measures of the game-based assessment tool would:

1. Exhibit high test retest reliability (Intra class correlations >0.7), and Standard error of measures less than 20% of the group mean.
2. Show moderate convergent validity (correlations, r>0.06) with the primary outcome measures.

RESEARCH PROJECT OBJECTIVE 2

An feasibility randomized clinical trial will be conducted to examine recruitment, acceptability, compliance and therapy dosage of the CRP program and to estimate the treatment effect of the repetitive task practice game-aided exercise program on dynamic balance skills, transfers from sitting to standing, turning, stepping, and gait function in children aged 3-8 years (n= 50) diagnosed with CP. Preliminary estimation of treatment effects and the calculation of effect size and sample size for a full scale definitive RCT will be determined on the basis of pre and post scores of the primary outcome measures. Two groups of children will be examined, one group will receive the experimental game-aided balance training program and the other group will receive usual conventional balance training program. Each program would take 12 weeks, three therapy sessions per week. Using a process of randomization, every child will be assigned to either experimental or control group after the initial assessment and screening. Before the treatment sessions begin, after the end of 12 weeks, a clinician will conduct regular assessment sessions with the participant to mark the progress till date.

The feasibility of assessment tool embedded in the game-aided rehabilitation platform and also the usability, safety and appeal of the protocol will be examined. An estimation of effectiveness on this sample using mixed method Analysis of Variance for within (repeated measure) and between group effects will be observed.

RESEARCH PROJECT OBJECTIVE 3

It is important to develop evidence on quality and actual dosage of an intervention to be delivered to create a positive outcome on the transfer of skills to functional performance. Thus during each session the dosage of intervention will be determined by recording the duration, intensity and quality of the balance and mobility exercises delivered with this treatment model at each session. In turn the aim is to develop a dose-response relationship for clinical use of this CRP program in rehabilitation of children with CP.

STUDY DESIGN: Feasibility Randomized Clinical Trial

METHOD OF COLLECTION OF DATA:

Ethical clearance for the study will be obtained from the Institutional Ethical Committee of S. D. M. College of Medical Sciences and Hospital, Dharwad. Participants will be recruited by clinicians working in Outpatient Department of Physiotherapy, S.D.M. Hospital, Dharwad, Karnataka, India. Parents of the participants will be approached for consent to take part in the study, the study participants in experimental group will be asked to sit or stand (as per the screening result) on fixed and compliant surfaces and to use objects instrumented with the miniature motion mouse to play various therapeutic yet entertaining games while handling and moving the test therapeutic objects using bi-manual grip gradually progressing to head rotations (with the mouse mounted on a cap worn by the participant) and finally using trunk movements as a part of experimental therapy protocol. The head movements and trunk movements will increase the body sway and hence increase the balance cost of the exercises to result in improvement in balance control. The speed and the amount of head or trunk movements (i.e. balanced costs) will be graded by adjusting the difficulty level of game play. While performing CGR the children will be standing on a thin pressure mat (placed over fixed or compliant surface). This will allow us to record the information of Center of Foot Pressure (COP) displacement [body sway] while game-aided balance training intervention implementation. This information will be used to quantify the intensity and duration of each exercise (i.e. therapy dose) for objective 3.

The following is a summary of the experimental balance training protocol:

1. Sitting Balance exercises while the child maintains sitting balance while playing the interactive computer games starting with bi-manual object placed in hands for controlling the games, then using the head rotation movements to control the games and then progressing to use of trunk motions to control games while balancing on the compliant surface (air bladder); in order to progress by increasing the balance costs.
2. Standing Balance exercises progressing from a fixed support surface to uneven and compliant support surfaces like progression from standing over ground then on sponge and then on air bladder as the child tolerates, i.e. increased balance costs.
3. Progression then to balancing while performing the visuomotor and visuospatial game tasks such as playing the games starting with bimanual object placed in hands for controlling the games, then using the head rotation movements to control the games and then progressing to use of trunk motions to control games while balancing on the compliant surface.
4. Progression to single-leg stance and to stepping activities. The control group participants will be receiving the conventional physical therapy protocol for balance rehabilitation.

The following is a summary of the conventional physical therapy balance training protocol:

1. Active-assisted stretching exercises for lower limb musculature focusing on postural control and improvement in dynamic stability,
2. Balance and weight bearing exercises with multi-directional reach outs associated with trunk movements on fixed surface gradually progressing to unstable movable and compliant surfaces,
3. Weight transfer exercises with multi-directional reach outs and
4. Stepping exercises in different directions on variety of surfaces.

Further if parents have any queries regarding the study can be reported to the principal investigators. The parents would be reassured that information would be kept confidential and will be used only for study purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Children with confirmed medical diagnosis of Cerebral Palsy
2. Age group - 3-8 years
3. GMFCS level - 1-3
4. Modified Ashworth scale level 0 to +1.

Exclusion criteria:

1. Visual or auditory impairment such that the interaction with the video games is difficult;
2. Secondary orthopedic complications due to neurodegenerative disease (NDD)
3. Modified Ashworth scale level > +1,
4. GMFCS level - 4-5,
5. Recent Botulinum toxin therapy (less than 6 months);
6. Recent Surgical intervention,
7. Cognitive impairment
8. Non willing parents,
9. Seizures, or
10. Complex communication disorders.

Tools for Screening:

1. Gross Motor Function Classification System (GMFCS) &
2. Modified Ashworth Scale.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scale-2 (PDMS-2) | Changes from baseline to post-intervention i.e. at 12 weeks
  The PDMS-2 is an early childhood motor development program that provides both in-depth assessment and training or remediation of gross and fine motor skills. The assessment is composed of six sub-tests that measure interrelated motor abilities that develop early in life. It is designed to assess the motor skills of children from birth through 5 years of age. The Stationary, Locomotion and Object Manipulation sub-tests of this scale will be used as the primary outcome measures of the study.
Gross Motor Function Measure | Changes from baseline to post-intervention i.e. at 12 weeks
  The GMFM is an observational clinical tool designed to evaluate change in gross motor function in children with CP aged between 5 months to 16 years. The sitting, crawling and kneeling, standing, walking and running components of the scale will be used as the primary outcome measures of the study.
COP Displacement Measures | Changes from baseline to post-intervention i.e. at 12 weeks
  The assessment of the center of foot pressure (COP) displacement using BodiTrack Pressure Mapping System while performance of the modified CTSIB tasks on normal and compliant surfaces will be taken at baseline and after implementation of intervention to assess the response of the balance control in variety of conditions.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - School of Medical Rehabilitation , University of Mantioba, Winnipeg, Manitoba
  - University of Manitoba, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No